CLINICAL TRIAL: NCT01444547
Title: A Phase Ⅱ Study on Low-expression and High-expression of ERCC1 in Recurrent or Metastastic Esophageal Cancer Patients Treated With Biweekly Paclitaxel and Cisplatin
Brief Title: A Study on Predictive Value of ERCC1 in Esophageal Cancer Patients Treated With Paclitaxel and Cisplatin
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Collaborators: Beijing Municipal Science & Technology Commission (Other)
Responsible Party: Principal Investigator, Jing Huang, Principle Investigator, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CH-GI-021; Z111107058811023 (Registry Identifier: CH-GI-021)
Record Dates: First submitted 2011-09-28; First posted 2011-09-30 (Estimated); Last update posted 2014-05-06 (Estimated); Status verified 2014-05

CONDITIONS: Esophageal Cancer
Keywords: esophageal cancer; paclitaxel; cisplatin
MeSH Terms: conditions — Esophageal Neoplasms | interventions — TP protocol; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- single-arm Paclitaxel-Cisplatin (Experimental)
  Interventions: Drug: paclitaxel and cisplatin

INTERVENTIONS:
Drug: paclitaxel and cisplatin — Paclitaxel 150 mg/m2 will be administered as an intravenous (IV) infusion over 3 hour on Days 1; Cisplatin 50 mg/m2 will be administered as an intravenous (IV) infusion on Days 2, and to take enough hydration in the day and the next day.
  14 days as a cycle, up to 8 cycles.
  Other Names: Paclitaxel,Beijing Union Pharmaceutical Factory

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of first-line chemotherapy with cisplatin and paclitaxel in esophageal cancer

DETAILED DESCRIPTION:
Open label single arm phase II study of cisplatin and paclitaxel in patients with recurrent or metastatic esophageal cancer. 92 Patients will be enrolled in this local trial. The primary objective of this study is to determine the response rate of the treatment.Schedule for this study is as follows: paclitaxel 150 mg/m2 will be administered as an intravenous infusion over 3 hour on Days 1, followed by cisplatin 50 mg/m2 on Days 2. This study will also include the investigation of ERCC1 expression in order to assess determinants of efficacy of the treatment with cisplatin and paclitaxel in the study population.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven diagnosis of the squamous cell carcinoma or adenocarcinoma of esophagus
* locally advanced, recurrent or metastatic disease
* Performance Status of 0-2 on the Eastern Cooperative Oncology Group (ECOG) performance status Scale
* Previous adjuvant or pre-operative chemotherapy without containing paclitaxel or platinum at least 12 months before enrollment
* Adequate organ function including the following:

Bone marrow: absolute neutrophil count (ANC) >or equal to 1.5 * 109/L, platelets >or equal to 100 *109/L, hemoglobin > or equal to 10 g/dL.

Hepatic: bilirubin < or equal to 1.5 x ULN; alkaline phosphatase, aspartate transaminase (AST) and alanine transaminase (ALT) < or equal to 3 x ULN (alkaline phosphatase, AST, ALT minor or equal to 5 x ULN is acceptable if liver has tumor involvement), serum albumin > or equal to3g/dL.

Renal: Calculated creatinine clearance major or equal to 60 ml/min (using the standard Cockcroft-Gault formula).

Exclusion Criteria:

* No Prior palliative chemotherapy for advanced disease
* Previous radiation therapy is allowed but should have been limited and must not have included whole pelvis radiation. Patients must have recovered from the toxic effects of the treatment prior to study enrollment (except for alopecia). Prior radiotherapy must be completed at least 30 days before study enrollment
* Known or suspected brain metastasis
* Second primary malignancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2007-01; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | 5 year
  The primary objective of this study is to determine the response rate of paclitaxel plus cisplatin as first-line therapy in patients with locally advanced, recurrent or metastatic esophageal carcinoma

SECONDARY OUTCOMES:
Time to event efficay | 5 year
  The following time to event efficacy measures:
  * Duration of overall response for responding patients
  * Time to documented progressive disease
  * Overall survival
  * The quantitative and qualitative toxicity of paclitaxel plus cisplatin.
  * Determinant of efficacy of the treatment with paclitaxel and cisplatin in the patient population by means of the analysis of ERCC1

CONTACTS AND LOCATIONS:
Overall Officials: Jing Huang, M.D.,Ph.D, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, China

REFERENCES:
- [Result] Lee S, Park YH, Kim KH, Cho EY, Ahn YC, Kim K, Shim YM, Ahn JS, Park K, Im YH. Thymidine synthase, thymidine phosphorylase, and excision repair cross-complementation group 1 expression as predictive markers of capecitabine plus cisplatin chemotherapy as first-line treatment for patients with advanced oesophageal squamous cell carcinoma. Br J Cancer. 2010 Sep 7;103(6):845-51. doi: 10.1038/sj.bjc.6605831. Epub 2010 Aug 10. PMID 20700125
- [Result] Olaussen KA, Fouret P, Kroemer G. ERCC1-specific immunostaining in non-small-cell lung cancer. N Engl J Med. 2007 Oct 11;357(15):1559-61. doi: 10.1056/NEJMc072007. No abstract available. PMID 17928611